CLINICAL TRIAL: NCT05473780
Title: Observational Study: Oxygen Therapy Monitoring in COPD Patients Using Connected Devices.
Brief Title: Oxygen Therapy Remote Monitoring in COPD Patients.
Status: Active, not recruiting | Type: Observational
Sponsor: Vivisol (Other)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Other Study IDs: O2 Connect; IDRCB 2022-A00825-38 (Other: French National Health Agency)
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: long term oxygen therapy; compliance; quality of life; exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background : Long-term oxygen therapy is prescribed for patients with severe COPD. The aim of oxygen therapy is to administer oxygen at a concentration level higher than that of ambient air, in order to treat or prevent the symptoms and manifestations of arterial hypoxemia; this therapy can be applied either in an acute situation or as a long-term treatment, in cases of stabilized severe chronic hypoxemia.

Currently, pneumologists do not have the possibility, between 2 consultations spaced several months apart, to measure the patient's compliance with the treatment (adherence to oxygen therapy) nor the respect of the prescribed dosage (O2 flow and duration). In addition to the patient's adherence to the treatment, the specialist does not have the possibility to assess the patient's physical activity (walking ...).

This observational study is a e-health, prospective, multicenter study conducted in France under the control of pneumologists.

The main objective of this study is to evaluate the adherence to oxygen therapy in real life, and its evolution, in COPD patients justifying a long term oxygen therapy in stable state.

DETAILED DESCRIPTION:
The observational study consists in collecting physiological data (cardiorespiratory and physical activity) and use of the oxygen therapy device in real life during the first months after the initiation of treatment.

For this purpose, two connected medical devices will be provided to each patient during 2 periods of 2 weeks (weeks 6 to 8 then weeks 12 to 14 after the initiation of oxygen therapy). The devices are: 1/ a connected watch that continuously measures vital parameters (heart rate and blood oxygen saturation), and physical activity parameters (no. of steps, distance, duration of effort), and 2/ a Teleox device that remotely monitors patients equipped with an oxygen source (it measures the oxygen flow rate requested by the patient, the duration of use of the oxygen source, and the breathing rate).

Study design: a cohort of 250 patients with COPD newly initiated a long term oxygen therapy will be enrolled in the study and follow-up over 6 months. Data will be collected by lung specialists and home health care provider teams at 2 months, 3.5 months and 6 months post-initiation of oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients who require the initiation of a long term oxygen therapy.
* Patient agreeing to use a connected watch and a TeleOx for the remote monitoring of their parameters and physical activity.
* Non-smoker, ex-smoker, or patient agreeing to stop smoking.
* Life expectancy greater than 6 months.
* Signed informed consent form,
* Subject affiliated to a health insurance system, or is a beneficiary.

Exclusion Criteria:

* Patient initiated on oxygen therapy prior to the inclusion visit.
* Patient with cognitive impairment.
* Simultaneous participation in a health intervention research,
* Vulnerable subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of COPD patients who initiate long-term oxygen therapy.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of compliance of long term oxygen therapy | 3.5 months
  For each patient, the average daily duration of oxygen use (expressed as numbers of hours of oxygen use per day) will be measured on period of 14 consecutive days at different times after the initiation of oxygen therapy (weeks 6 to 8, and then weeks 12 to 14). The duration of oxygen use is measured using the TeleOx medical device placed in each oxygen source (fixed and portable sources).

SECONDARY OUTCOMES:
Impact of long term oxygen therapy on heart rate | Month 2, Month 3.5
  For each patient, the average and maximum daily heart rate (expressed as beats/minute) will be measured on period of 14 consecutive days at different times after the initiation of oxygen therapy (weeks 6 to 8, and then weeks 12 to 14). The heart rate is measured by the connected watch all along the day.
Impact of long term oxygen therapy on oxygen saturation in the blood (SpO2) | Month 2, Month 3.5
  For each patient, the average nightime and daytime SpO2 (expressed in %) will be calculated by period of 14 consecutive days at different times after the initiation of oxygen therapy (weeks 6 to 8, and then weeks 12 to 14). The SpO2 is measured by the connected watch (automatically at night and manually in day).
Impact of long term oxygen therapy on the respiratory rate | Month 2, Month 3.5
  For each patient, the median, maximum, and 95th percentile daily respiratory rate (expressed in cycles/minute) will be measured on period of 14 consecutive days at different times after the initiation of oxygen therapy (weeks 6 to 8, and then weeks 12 to 14). The respiratory rate is measured using the TeleOx medical device placed in each oxygen source (fixed and portable sources).
Impact of long term oxygen therapy on the physical activity in terms of duration of effort | Month 2, Month 3.5
  For each patient, the total duration of effort per day (expressed in hours) will be measured on period of 14 consecutive days at different times after the initiation of oxygen therapy (weeks 6 to 8, and then weeks 12 to 14). The total duration of effort is measured by the connected watch.
Impact of long term oxygen therapy on the physical activity in terms of duration of number of steps | Month 2, Month 3.5
  For each patient, the total number of steps per day will be measured on period of 14 consecutive days at different times after the initiation of oxygen therapy (weeks 6 to 8, and then weeks 12 to 14). The number of steps is measured by the connected watch.
Impact of long term oxygen therapy on the health related quality of life of COPD patients | At oxygen therapy initiation (baseline), Month 2, Month 3.5
  The quality of life will be assessed using the COPD-specific health related quality of life questionnaire named VQ11.
  The questionnaire VQ11 comprises 11 items distributed across three components (functional: 3 items, psychological: 4 items, social: 4 items). The global score ranges from 11 to 55 points; higher scores mean a better quality of life.
Impact of long term oxygen therapy on the respiratory function | At inclusion, Month 6
  The pulmonologist will assess the evolution of respiratory function according to good medical practice with the pulmonary functional tests. Based on the VEMS/CV value (expressed in %), the pulmonologist judges if the prescribed long term oxygen therapy is sufficient to normalize the respiratory function or if the treatment must be modified.
Assessment of exacerbation | Month 6
  The pulmonologist will assess the number of exacerbation that occured during the first 6-months of long term oxygen therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ari CHAOUAT, Pr, Principal Investigator — CHRU Nancy-Université de Lorraine
Locations (36):
- France (36):
  - CHIAP, Aix-en-Provence
  - CH Nord Ardèche, Annonay
  - Cabinet privé, Antibes
  - Hopital Privé de La Casamance, Aubagne
  - Cabinet libéral, Avignon
  - CH Avignon, Avignon
  - CH Blois, Blois
  - CH Bligny, Briis-sous-Forges
  - CH Cannes, Cannes
  - Hôpital Percy, Clamart
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CH Draguignan, Draguignan
  - Cabinet libéral, Foix
  - CH Emile Roux, Le Puy-en-Velay
  - Cabinet libéral, Le Puy-en-Velay
  - CH Libourne, Libourne
  - Hôpital La Louvière, Lille
  - Centre médical Parot, Lyon
  - Hôpital Saint Joseph, Marseille
  - Hôpital d'Instruction des Armées Laveran, Marseille
  - AP-HM Hopital nord, Marseille
  - CH de Martigues, Martigues
  - GHSIF / CH Melun, Melun
  - GHI Le Raincy, Montfermeil
  - CHRU Nancy-Université de Lorraine, Nancy
  - Polyclinique des fleurs, Ollioules
  - CH Louis Giorgi d'Orange, Orange
  - CH de Perpignan, Perpignan
  - Pneumology practice, Perpignan
  - CHU de Bordeaux, Pessac
  - Cabinet libéral, Poissy
  - CH St Nazaire, Saint-Nazaire
  - MGEN, Sainte-Feyre
  - cabinet du dr Radu Horia Bumbea, Sallanches
  - Cabinet de Pneumologie, Toulon
  - Clinique Pasteur, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided